CLINICAL TRIAL: NCT05403281
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of Fixed-dose Combination of DW6012 and Loose-combination of Each Component in Healthy Adult Volunteers
Brief Title: A Pharmacokinetic Study of DW6012 (FDC of Dapagliflozin and Sitagliptin) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW6012-I-1
Record Dates: First submitted 2022-05-04; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Healthy Subjects
Keywords: Dapagliflozin; Sitagliptin; sitagliptin phosphate; Dapagliflozin propanediol
MeSH Terms: interventions — dapagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: Dapagliflozin and Sitagliptin / Period 2: DW6012
  Interventions: Drug: DW6012
- Sequence B (Experimental): Period 1: DW6012/ Period 2: Dapagliflozin and Sitagliptin
  Interventions: Drug: DW6012

INTERVENTIONS:
Drug: DW6012 — Drug: DW6012 Single oral administration of DW6012 after an overnight fast
  Drug: Dapagliflozin and Sitagliptin Single oral administration of Dapagliflozin and Sitagliptin after an overnight fast
  Other Names: Dapagliflozin and Sitagliptin

SUMMARY:
This study is to compare and evaluate the safety and pharmacokinetic characteristics (PK) after administration of DW6012 and each component in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged up to 19 years
* Subjects weighing at least 50.0 kg and no more than 100 kg (inclusive) with a BMI between 18.5 kg/m2 and 30.0 kg/m2
* Subjects with neither congenital nor chronic diseases requiring treatment, and no abnormal symptoms or findings upon medical examination
* Subjects considered eligible for the study participation in accordance to the results of clinical laboratory tests, vital signs, physical examinations and 12-lead ECG conducted at the time of screening, based on the investigational product (IP) characteristics
* Subjects who has a full understanding in participation of the study, voluntarily provide a written consent in participation, and give full agreement in following the subject guidelines throughout the entire study period

Exclusion Criteria:

* Subjects with any clinically significant hepatic, renal, nervous, respiratory, endocrine, circulatory, tumor, genitourinary, cardiovascular, digestive, musculoskeletal systemic diseases or other medical history
* Subjects with genetic problems such as Lapp lactase deficiency (Lapp) or galactose intolerant galactose due to galactose intolerance
* Subjects with a past medical history of gastrointestinal disease or gastrointestinal surgeries which may affect the absorption, distribution, metabolism and excretion of the IP
* Pregnant subjects with a positive urine HCG test, or lactating female subjects
* Subjects with hypersensitivity reactions or a clinically significant medical history of hypersensitivity reactions to drug substances and additives containing drug substances or other drugs
* Subjects with clinically significant 12-lead ECG findings at the time of screening
* Subjects with clinically significant laboratory test results as follows: Liver function test (AST, ALT, ALP, γ-GTP and total bilirubin), Creatinine, eGFR
* Subjects with a past history of drug abuse or a positive urine drug test
* Subjects with SBP ≥ 150 mmHg or ≤ 90 mmHg; DBP ≥ 100 mmHg or ≤ 60 mmHg; PR ≤ 40 bpm or ≥ 100 bpm at the time of screening
* Subjects following an unusual diet or consumption of food which may affect the absorption, distribution, metabolism and excretion of the IP
* Subjects who have administered any prescription drugs or herbal medicines that may affect the characteristics of clinical investigational drugs within 2 weeks prior to the first administration date, or have administered any over-the-counter (OTC) or vitamin preparations within 10 days
* Subjects taking drugs known to significantly induce or inhibit drug metabolizing enzymes, including barbitals within 1 months prior to the first IP administration
* Subjects who have participated and were given any other study drugs in other clinical study within 6 months prior to the first IP administration
* Subjects who have consistently drunk alcohol within 6 months
* Subjects who have smoked more than 10 cigarettes/day on average
* Subjects who have eaten or cannot refrain from eating grapefruit (grapefruit)-containing food from 48 hours before the first administration until the time of PSV
* Subjects who have consumed or cannot refrain from consuming caffeine-containing food during the period from 24 hours prior to administration of each period to the time of the last blood sampling
* Subjects who have done and are unable to refrain from strenuous activity
* Subjects who are planning for pregnancy or not willing to use a medically reliable forms of contraception
* Subjects otherwise considered ineligible for participation due to other reasons including clinical laboratory test results not mentioned in the inclusion/exclusion criteria at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
AUC0-t of Dapagliflozin and Sitagliptin | up to 48 hours
Cmax of Dapagliflozin and Sitagliptin | up to 48 hours

SECONDARY OUTCOMES:
AUCinf | up to 48 hours
Tmax | up to 48 hours
t1/2 | up to 48 hours
CL/F | up to 48 hours
Vd/F | up to 48 hours
AUCextra | up to 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No